CLINICAL TRIAL: NCT02870296
Title: Anticoagulation Medical Home for High-Risk Patients With Venous Thromboembolism: Patient Education, Anticoagulant Decision-Making, and Patient Self-Efficacy in the Home Coordinated by the UMass Anticoagulation Team
Brief Title: Anticoagulation Medical Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Alok Kapoor, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00010242
Record Dates: First submitted 2016-06-10; First posted 2016-08-17 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Venous Thromboembolism; Patient-Centered Care
MeSH Terms: conditions — Venous Thromboembolism | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive usual care; no interventions will be administered.
- Intervention (Experimental): Interventions will be administered to this group. Patients in the Intervention Group will: 1) have an in-home pharmacist medication assessment; 2) receive enhanced medication instructions (including pictograms); 3) receive an additional individualized assessment and educational session with a clinician provider related to the medication management for their disease (VTE).
  Interventions: Behavioral: Enhanced Assessment and Education

INTERVENTIONS:
Behavioral: Enhanced Assessment and Education — Patients in the Intervention Group will: 1) have an in-home pharmacist medication assessment; 2) receive enhanced medication instructions (including pictograms); 3) receive an additional individualized assessment and educational session with a clinician provider related to the medication management for their disease (VTE).
  Arms: Intervention

SUMMARY:
The primary study goal is to improve the quality of care transitions for patients with new episodes of venous thromboembolism (VTE).

Primary Outcomes: To measure differences in the quality of care transition, as measured by the Care Transition Measure (CTM)-15 in the investigators target population of patients with incident VTE randomized to either a multicomponent, anticoagulation medical home intervention or usual care.

Secondary Major Outcomes: To measure the difference in recurrent VTE, major hemorrhage, all-cause re-admissions, and mortality between the investigators intervention and comparison groups at 30 and 90 days in the investigators target population.

Secondary Other Outcomes: To measure patient knowledge, health-related quality of life, and time in the therapeutic range (TTR) for patients on warfarin in the investigators target population.

ELIGIBILITY:
Inclusion Criteria:

* hospital admission;
* diagnosis of:

  * VTE (first or subsequent episode); or
  * DVT of leg or pelvis or upper extremities or other site confirmed by ultrasound or CT scan; or
  * PE with a positive CT spiral exam, pulmonary arteriogram, CT angiogram, or high probability ventilation perfusion scan.
* for whom it is anticipated the treating medical team will prescribe an oral anticoagulant upon hospital discharge.

Exclusion Criteria:

* Not engaged in Primary Care (has not seen a Primary Care Practitioner within the previous 18 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Care Transition Measure (CTM-15) | 30 days post hospital discharge
  15 item measure; measures 4 aspects of quality of transitional care

SECONDARY OUTCOMES:
Clinical Outcome: VTE Recurrence | 30 and 90 days post hospital discharge
  Measure the difference in recurrent VTE between intervention and comparison groups.
Clinical Outcome: Major Hemorrhage (noted in Medical Record and/or via patient self-report) | 30 and 90 days post hospital discharge
  Measure the difference in major hemorrhage between intervention and comparison groups- ISTH 2005 medical definition 14 - 2 unit drop in hemoglobin, 2 unit transfusion, or critical site bleed.
  - ISTH 2009 surgical definition 15 - surgical site 2 unit drop or 2 unit transfusion with increase in LOS, hemodynamic compromise, delay in rehab.
Clinical Outcome: Hospital Readmission (any unplanned hospital admissions noted in Medical Record and/or via patient self-report) | 30 and 90 days post hospital discharge
  Measure the difference between all cause hospital readmission (post-diagnosis of VTE) between intervention and comparison groups.
Clinical Outcome: Mortality | 30 and 90 days post hospital discharge
  Measure the difference in mortality between intervention and comparison groups.
Other Measure: Patient Knowledge (via questionnaire developed by Mazor et. al. 2007 Patient Educ Counsel and via investigator developed items) | 30 and 90 days post hospital discharge
  Measure patient knowledge and attitudes Mazor KM, Baril J, Dugan E, Spencer F, Burgwinkle P, Gurwitz JH. Patient education about anticoagulant medication: is narrative evidence or statistical evidence more effective? Patient Educ Couns. 2007 Dec;69(1-3):145-57. Epub 2007 Oct 17.
Other Measure: Quality of Life (VEINES-QOL/Sym questionnaire or PEmb-QoL questionnaire) | 30 and 90 days post hospital discharge
  Measure health-related quality of life for patients on warfarin and time in the therapeutic range (TTR) in our target population

CONTACTS AND LOCATIONS:
Overall Officials: Alok Kapoor, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Kapoor A, Bloomstone S, Javed S, Silva M, Lynch A, Yogaratnam D, Carlone B, Springer K, Maheswaran A, Chen X, Nagy A, Elhag R, Markaddy E, Aungst T, Bartlett D, Houng D, Darling C, McManus D, Herzig SJ, Barton B, Mazor K. Reducing Hospitalizations and Emergency Department Visits in Patients With Venous Thromboembolism Using a Multicomponent Care Transition Intervention. Inquiry. 2020 Jan-Dec;57:46958019900080. doi: 10.1177/0046958019900080. PMID 31965873
- [Derived] Kapoor A, Landyn V, Wagner J, Burgwinkle P, Huang W, Gore J, Spencer FA, Goldberg R, McManus DD, Darling C, Boudreaux E, Barton B, Mazor KM. Supplying Pharmacist Home Visit and Anticoagulation Professional Consultation During Transition of Care for Patients With Venous Thromboembolism. J Patient Saf. 2020 Dec;16(4):e367-e375. doi: 10.1097/PTS.0000000000000571. PMID 30702452